CLINICAL TRIAL: NCT04036578
Title: Efficacy of Pelvic Floor Muscle Training Using Bio-assisted Surface Electromyography in Women With Pelvic Floor Dysfunction With and Without Pelvic Organ Prolapse
Brief Title: Efficacy of Biofeedback in Women With Pelvic Floor Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 104145-F
Record Dates: First submitted 2019-05-03; First posted 2019-07-30 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2015-11

CONDITIONS: Pelvic Floor Dysfunction
Keywords: pelvic floor dysfunction; pelvic floor muscle training; pelvic organ prolapse; surface electromyographic program
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Intervention Model Description: A 12-week PFMT bio-assisted surface electromyographic program in group 1(Pelvic Floor Dysfunction Without POP Stage I~II) and group 2(Pelvic Floor Dysfunction With POP Stage I~II)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pelvic Floor Dysfunction With and Without POP (Other): group 1(Pelvic Floor Dysfunction Without POP Stage I~II) and group 2(Pelvic Floor Dysfunction With POP Stage I~II)
  Interventions: Device: A 12-week PFMT bio-assisted surface electromyographic program

INTERVENTIONS:
Device: A 12-week PFMT bio-assisted surface electromyographic program

SUMMARY:
Recent studies have found that pelvic floor muscle training can relieve pelvic organ prolapse related symptoms. However, the rate of cure or improvement of symptoms with exercise prescription, different compliance of the patient's behavior have great differences. Biofeedback is an instrument used to record the biological signals ( electrical activity) during a voluntary pelvic floor muscle contraction and provide feedback in auditory or visual form (a louder sound with a stronger squeeze or an increasing number of lights on a visual display as the strength of the squeeze increased). Therefore, this study would explore the efficacy of biofeedback-assisted pelvic floor muscle training in women with pelvic floor dysfunction with or without organ prolapse.

DETAILED DESCRIPTION:
Treatment options for pelvic floor dysfunction (PFD) vary depending on symptom severity. Conservative approaches such as pelvic floor muscle (PFM) exercises, biofeedback, and lifestyle advice are usually suggested for urgency incontinence (UI), overactive bladder (OAB), and mild-to-moderate pelvic organ prolapse (POP). Conservative management remains the gold standard of treatment for female UI and OAB. There is Level 1, Grade A evidence supporting pelvic floor muscle training (PFMT) as an effective treatment for UI and OAB, and Grade B evidence that pelvic floor muscle training (PFMT) reduces the symptoms of urogenital prolapse, although topographic changes are not expected. Most of the past literatures focused on the effectiveness of PFMT on single disease, but seldom explored its effectiveness on complex disease (i.e. women presenting with more than one type of PFD). In the real world, some degree of POP was present in 41% to 50% of women on physical examination, but only 3% of patients reported symptoms such as bearing down sensation of vagina. Besides, there was a number of studies that assessed the efficacy of PFMT as a treatment for women with POP, but rarely explored its effectiveness in both subjective and objective (anatomic) improvement of prolapse severity.

Biofeedback provides positive reinforcement to patients performing PFMT, therefore improves the quality of life of women with PFD. It can be achieved via several methods, including electromyography (EMG), manometry, or ultrasonography. A systematic review confirmed the benefit of adding of biofeedback to PFMT, but it was not clear whether this was the effect was related to another variable, such as the amount of health professional contact rather than the biofeedback.

ELIGIBILITY:
Inclusion Criteria:

1. pelvic organ prolapse for more than 3 months
2. more then 20 year old,less then 85 year old and acceptable to receive vaginal examination
3. need to match schedule with the investigator's clinic for 5 times,followed by individual therapy, each takes about 30 to 60 minutes, a total of 12 weeks of pelvic floor muscle exercises

Exclusion Criteria:

1. women who were unable to contract their PFMs due to cognitive deficit
2. had a neurological disorder
3. pregnant

Ages: 20 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2018-01-24 (Actual); Study Completion 2018-11-02 (Actual)

PRIMARY OUTCOMES:
electromyographic activity | Change from Baseline Electromyographic activity of the pelvic floor muscles (PFMs) and the synergistic abdominal muscles (SAMs) at 0,2,4,8,12 week
  Electromyographic activity of the pelvic floor muscles (PFMs) and the synergistic abdominal muscles (SAMs) during each session of PFMT(µV)
prolapse severity | Change from Baseline prolapse severity with subjectively and objectively (using the POP Quantification System) at 12 week
  The prolapse severity was assessed subjectively and objectively (using the POP Quantification System) before and after the intervention in women with POP.